CLINICAL TRIAL: NCT05468710
Title: The Prognostic and Predictive Role of Inflammatory Blood Markers in Early and Locally Advanced Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Brief Title: Inflammatory Blood Markers in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tawfik Helmy, clinical oncology assistant lecturer, faculty of medicine, Ain Shams University
Other Study IDs: MD 134/2022
Record Dates: First submitted 2022-07-14; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most threatening disease in women. Neoadjuvant chemotherapy is a commonly used for the treatment. Inflammation plays an important role in tumor proliferation, metastasis, and resistance to chemotherapy. Inflammatory blood markers (IBM) reflect the balance between host inflammatory and immune status. Different IBM have been reported as prognostic factors for survival and predictive factors for pathological complete response and toxicity. Our aim to evaluate these IBM in breast cancer patients receiving neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Inflammation, recognized as one of the 10 hallmarks of cancer (seventh hallmark of cancer), contributes to tumour proliferation, angiogenesis, metastasis, and resistance to chemotherapy. In general, white blood cell count reflects an individual's systemic and/or local inflammatory status. Neutrophils are known to regulate the tumour microenvironment and produce cytokines, chemokines, and growth factors that may promote angiogenesis as well as tumour cell proliferation and migration. The M2 phenotype tumour-associated macrophages (TAMs) deriving from circulating monocytes exist within the tumour microenvironment and promote metastasis and immunosuppression. It was reported that peripheral monocyte count was associated with the density of the TAMs, and high absolute monocyte count predicted poor survival in cancer patients. Platelets are other cells contributing to cancer-favoured inflammation by various mechanisms. For example, the activated platelets inhibit the interaction between tumour cells and cytolytic immune cells by forming a layer around tumour cells and support tumour growth via the secretion of several factors such as TGF-β. Hence, high platelet counts were reported to be associated with adverse outcomes in breast cancer. In contrast, lymphocytes are responsible for antitumor-specific immune response including T-lymphocyte tumour infiltration and cytotoxic T-lymphocyte-mediated antitumor activity.

Inflammatory blood markers (IBM) have emerged as potential prognostic factors for survival in different types of cancers including breast cancer, as well as predictive factors for histological response after neo-adjuvant chemotherapy. IBM include leucocyte count, lymphocyte count, neutrophil count, and ratios such as platelet to lymphocyte ratio (PLR) or neutrophil to lymphocyte ratio (NLR), and monocyte to lymphocyte ratio (MLR). Starting from these findings, NLR, MLR, and PLR, indices reflecting the balance between inflammation and immunoreaction in cancer, were reported to have predictive value in NAC response in many breast cancer studies.

There are conflicting reports about which index provides the best prediction for the efficacy of NAC in breast cancer. For example, Eren et al. reported that NLR was the only independent predictive factor of pathological complete response (pCR) among blood-derived inflammation markers in multivariate analysis. In another study conducted by Peng et al., multivariate analysis of 808 breast cancer patients showed that the lymphocyte-monocyte ratio was the only independent predictive factor for the efficacy of NAC among these inflammatory markers. In addition, Hu et al. stated that PLR had superior efficacy to NLR in predicting NAC response.

Different studies tried to integrate different peripheral blood immune cells as, Jiang et al., that used systemic immune-inflammation index (SII); is based on neutrophil (N), platelet (P) and lymphocyte (L) counts, and stated that prognostic utility of (SII) was superior to that of NLR and PLR. Also Dong et al used the systemic inflammation response index (SIRI); an integrated indicator based on the counts of peripheral venous blood neutrophils(N), monocytes(M) and lymphocytes(L), and stated the prognostic value of the (SIRI) for pCR was superior to that of NLR.

Pan-Immune-Inflammation-Value (PIV) is a new blood-based biomarker integrating different peripheral blood immune cell subpopulations-neutrophil, platelet, monocyte, and lymphocyte. Due to its potential to represent comprehensively patient's immunity and systemic inflammation, PIV was proposed as a stronger predictor of outcomes in cancer patients receiving cytotoxic chemotherapy, immunotherapy, and targeted therapy. Recently, Ligorio reported that PIV was firmly associated with survival and outperformed NLR, PLR, and MLR in predicting survival in patients with HER-2 positive advanced breast cancer.

Sahin et al., stated that pre-treatment PIV seems as a predictor for pCR and survival, outperforming NLR, MLR, PLR in Turkish women with breast cancer who received NAC.

Some studies stated that the SIRI and SII had no significance on toxicities like peripheral neuropathy and neutropenia. However, other studies reported NLR as predictive factor for febrile neutropenia.

These integrated indicators may fully reflect the balance between host inflammatory and immune status compared with NLR, MLR and PLR and other conventional haematological parameters.

These conflicting results have raised the need for a study to evaluate these inflammatory blood markers in patients with breast cancer receiving neo adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or more.
* Histologically proven invasive breast cancer.
* Above cT1 stage, any N Stage with no distant metastasis M0.
* All subtypes are included, either HR (ER, PR) positive or negative, HER2 positive or negative.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2.
* Patients who completed their systemic neoadjuvant therapy.
* Available baseline complete blood picture before starting treatment.

Exclusion Criteria:

* Second malignancy.
* Patients with early breast cancer cT1 (≤ 2 cm) N0.
* Metastatic patients M1.
* Patients with systemic inflammatory diseases or autoimmune diseases (Type I Diabetes mellitus, Systemic Lupus Erytheromatosis, Rheumatoid Arthritis, Sjogren's syndrome, Behcet disease).
* Pregnancy-related breast cancer.
* Patients with chronic diseases (liver cirrhosis, or end-stage renal disease).
* Patients on systemic steroids as well as those under NSAIDS or other immunomodulators (as Methotraxate, Tacrolimus and Cyclosporine).
* Patient who received radiotherapy or endocrine or targeted therapy prior to neoadjuvant chemotherapy.
* Patients who started but didn't complete neoadjuvant systemic therapy.
* Patients who didn't undergo surgery after neoadjuvant systemic therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasive breast cancer, Above cT1 stage, all subtypes are included, who completed neoadjuvant systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between inflammatory blood marker (neutrophil to lymphocyte ration (NLR)) and rate of pathological complete response (PCR), and neutropenia / peripheral neuropathy (CTCAE grade). | 1 year
  * The neutrophil to lymphocyte ratio (NLR) was provided by the ratio between the absolute count of neutrophils and the absolute count of lymphocytes (NLR = N /L)
  * Pathological complete response (PCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system).
  * Toxicity endpoint, will be retrieved and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Correlation between inflammatory blood marker (Platelet to lymphocyte ratio(PLR)) and rate of pathological complete response (PCR), and neutropenia / peripheral neuropathy (CTCAE grade). | 1 year
  * The Platelet to lymphocyte ratio(PLR) was provided by the ratio between the absolute count of platelets and the absolute count of lymphocytes (PLR= P/L)
  * Pathological complete response (PCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system).
  * Toxicity endpoint, will be retrieved and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Correlation between inflammatory blood marker (monocyte to lymphocyte ratio(MLR)) and rate of pathological complete response (PCR), and neutropenia / peripheral neuropathy (CTCAE grade). | 1 year
  * The Monocyte to lymphocyte ratio (MLR) was provided by the ratio between the absolute count of monocytes and the absolute count of lymphocytes (MLR= M/L)
  * Pathological complete response (PCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system).
  * Toxicity endpoint, will be retrieved and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Correlation between inflammatory blood marker (systemic immune-inflammation index(SII)) and rate of pathological complete response (PCR), and neutropenia / peripheral neuropathy (CTCAE grade). | 1 year
  * The systemic immune-inflammation index is based on neutrophil (N), platelet (P) and lymphocyte (L) counts (SII = N × P/L) .
  * Pathological complete response (PCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system).
  * Toxicity endpoint, will be retrieved and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Correlation between inflammatory blood marker (systemic inflammation response index (SIRI)) and rate of pathological complete response (PCR), and neutropenia / peripheral neuropathy (CTCAE grade). | 1 year
  * systemic inflammation response index (SIRI) is based on neutrophils(N), monocytes(M) and lymphocytes(L) (SIRI=N×M/L) .
  * Pathological complete response (PCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system).
  * Toxicity endpoint, will be retrieved and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Correlation between inflammatory blood marker (Pan-Immune-Inflammation-Value (PIV)) and rate of pathological complete response (PCR), and neutropenia / peripheral neuropathy (CTCAE grade). | 1 year
  * Pan-Immune-Inflammation-Value (PIV) is based on neutrophils(N), monocytes(M),platelet(P) and lymphocytes(L) (PIV=N×M×P/L).
  * Pathological complete response (PCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system).
  * Toxicity endpoint, will be retrieved and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Correlation between inflammatory blood marker (neutrophil to lymphocyte ration (NLR)) and disease-free survival (DFS) and overall survival (OS). | 1 year
  * The neutrophil to lymphocyte ratio (NLR) was provided by the ratio between the absolute count of neutrophils and the absolute count of lymphocytes (NLR = N /L)
  * Disease free survival (DFS) is defined as the time from diagnosis to the date of relapse (local recurrence or metastases to distant sites) and/or death from any cause.
  * Overall survival (OS) is defined from the date of diagnosis to the date of death or the end of follow-up.
Correlation between inflammatory blood marker (Platelet to lymphocyte ratio(PLR)) and disease-free survival (DFS) and overall survival (OS). | 1 year
  * The Platelet to lymphocyte ratio(PLR) was provided by the ratio between the absolute count of platelets and the absolute count of lymphocytes (PLR= P/L)
  * Disease free survival (DFS) is defined as the time from diagnosis to the date of relapse (local recurrence or metastases to distant sites) and/or death from any cause.
  * Overall survival (OS) is defined from the date of diagnosis to the date of death or the end of follow-up.
Correlation between inflammatory blood marker ( Monocyte to lymphocyte ratio (MLR)) and disease-free survival (DFS) and overall survival (OS). | 1 year
  * The Monocyte to lymphocyte ratio (MLR) was provided by the ratio between the absolute count of monocytes and the absolute count of lymphocytes (MLR= M/L)
  * Disease free survival (DFS) is defined as the time from diagnosis to the date of relapse (local recurrence or metastases to distant sites) and/or death from any cause.
  * Overall survival (OS) is defined from the date of diagnosis to the date of death or the end of follow-up.
Correlation between inflammatory blood marker (Systemic immune-inflammation index (SII)) and disease-free survival (DFS) and overall survival (OS). | 1 year
  * The systemic immune-inflammation index (SII) is based on neutrophil (N), platelet (P) and lymphocyte (L) counts (SII = N × P/L) .
  * Disease free survival (DFS) is defined as the time from diagnosis to the date of relapse (local recurrence or metastases to distant sites) and/or death from any cause.
  * Overall survival (OS) is defined from the date of diagnosis to the date of death or the end of follow-up.
Correlation between inflammatory blood marker (systemic inflammation response index (SIRI)) and disease-free survival (DFS) and overall survival (OS). | 1 year
  * systemic inflammation response index (SIRI) is based on neutrophils(N), monocytes(M) and lymphocytes(L) (SIRI=N×M/L) .
  * Disease free survival (DFS) is defined as the time from diagnosis to the date of relapse (local recurrence or metastases to distant sites) and/or death from any cause.
  * Overall survival (OS) is defined from the date of diagnosis to the date of death or the end of follow-up.
Correlation between inflammatory blood marker (Pan-Immune-Inflammation-Value (PIV)) and disease-free survival (DFS) and overall survival (OS). | 1 year
  * Pan-Immune-Inflammation-Value (PIV) is based on neutrophils(N), monocytes(M),platelet(P) and lymphocytes(L) (PIV=N×M×P/L).
  * Disease free survival (DFS) is defined as the time from diagnosis to the date of relapse (local recurrence or metastases to distant sites) and/or death from any cause.
  * Overall survival (OS) is defined from the date of diagnosis to the date of death or the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nivine M Gado, phd, Study Director — Ain Shams University

REFERENCES:
- [Background] Sahin AB, Cubukcu E, Ocak B, Deligonul A, Oyucu Orhan S, Tolunay S, Gokgoz MS, Cetintas S, Yarbas G, Senol K, Goktug MR, Yanasma ZB, Hasanzade U, Evrensel T. Low pan-immune-inflammation-value predicts better chemotherapy response and survival in breast cancer patients treated with neoadjuvant chemotherapy. Sci Rep. 2021 Jul 19;11(1):14662. doi: 10.1038/s41598-021-94184-7. PMID 34282214
- [Background] Chen L, Kong X, Wang Z, Wang X, Fang Y, Wang J. Pre-treatment systemic immune-inflammation index is a useful prognostic indicator in patients with breast cancer undergoing neoadjuvant chemotherapy. J Cell Mol Med. 2020 Mar;24(5):2993-3021. doi: 10.1111/jcmm.14934. Epub 2020 Jan 27. PMID 31989747
- [Background] Corbeau I, Thezenas S, Maran-Gonzalez A, Colombo PE, Jacot W, Guiu S. Inflammatory Blood Markers as Prognostic and Predictive Factors in Early Breast Cancer Patients Receiving Neoadjuvant Chemotherapy. Cancers (Basel). 2020 Sep 18;12(9):2666. doi: 10.3390/cancers12092666. PMID 32962003
- [Background] Dong J, Sun Q, Pan Y, Lu N, Han X, Zhou Q. Pretreatment systemic inflammation response index is predictive of pathological complete response in patients with breast cancer receiving neoadjuvant chemotherapy. BMC Cancer. 2021 Jun 14;21(1):700. doi: 10.1186/s12885-021-08458-4. PMID 34126950
- [Background] Eren T, Karacin C, Ucar G, Ergun Y, Yazici O, Imamoglu GI, Ozdemir N. Correlation between peripheral blood inflammatory indicators and pathologic complete response to neoadjuvant chemotherapy in locally advanced breast cancer patients. Medicine (Baltimore). 2020 May 29;99(22):e20346. doi: 10.1097/MD.0000000000020346. PMID 32481414
- [Background] Hu Y, Wang S, Ding N, Li N, Huang J, Xiao Z. Platelet/Lymphocyte Ratio Is Superior to Neutrophil/Lymphocyte Ratio as a Predictor of Chemotherapy Response and Disease-free Survival in Luminal B-like (HER2-) Breast Cancer. Clin Breast Cancer. 2020 Aug;20(4):e403-e409. doi: 10.1016/j.clbc.2020.01.008. Epub 2020 Jan 30. PMID 32201163
- [Background] Jiang C, Lu Y, Zhang S, Huang Y. Systemic Immune-Inflammation Index Is Superior to Neutrophil to Lymphocyte Ratio in Prognostic Assessment of Breast Cancer Patients Undergoing Neoadjuvant Chemotherapy. Biomed Res Int. 2020 Dec 18;2020:7961568. doi: 10.1155/2020/7961568. eCollection 2020. PMID 33381583
- [Background] Ligorio F, Fuca G, Zattarin E, Lobefaro R, Zambelli L, Leporati R, Rea C, Mariani G, Bianchi GV, Capri G, de Braud F, Vernieri C. The Pan-Immune-Inflammation-Value Predicts the Survival of Patients with Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced Breast Cancer Treated with First-Line Taxane-Trastuzumab-Pertuzumab. Cancers (Basel). 2021 Apr 19;13(8):1964. doi: 10.3390/cancers13081964. PMID 33921727
- [Background] Peng Y, Chen R, Qu F, Ye Y, Fu Y, Tang Z, Wang Y, Zong B, Yu H, Luo F, Liu S. Low pretreatment lymphocyte/monocyte ratio is associated with the better efficacy of neoadjuvant chemotherapy in breast cancer patients. Cancer Biol Ther. 2020;21(2):189-196. doi: 10.1080/15384047.2019.1680057. Epub 2019 Nov 4. PMID 31684807